CLINICAL TRIAL: NCT01193270
Title: Single-Dose Vitamin E for Prevention of Mortality and Morbidity in Extremely Preterm Infants: Pilot Study
Brief Title: Vitamin E for Extremely Preterm Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NICHD-NRN-0044; U10HD021364 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027856 (NIH); U10HD027871 (NIH); U10HD027880 (NIH); U10HD027904 (NIH); U10HD034216 (NIH); U10HD036790 (NIH); U10HD040492 (NIH); U10HD040689 (NIH); U10HD053089 (NIH); U10HD053109 (NIH); U10HD053119 (NIH); U10HD053124 (NIH); UL1RR024139 (NIH); UL1RR024979 (NIH); UL1RR025744 (NIH); UL1RR025008 (NIH); UL1RR025761 (NIH); UL1RR025764 (NIH)
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Infant, Newborn; Infant, Small for Gestational Age; Infant, Very Low Birth Weight; Infant, Premature; Intracranial Hemorrhages
Keywords: NICHD Neonatal Research Network; Intraventricular Hemorrhage (IVH); Very Low Birth Weight (VLBW); Extremely Low Birth Weight (ELBW); Prematurity
MeSH Terms: conditions — Premature Birth; Intracranial Hemorrhages | interventions — Vitamin E; Tocopherols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin E (Experimental): A single intragastric dose of dl-α-tocopheryl acetate (Aquasol E®) 50 IU/kg.
  Interventions: Drug: Vitamin E
- Placebo (Placebo Comparator): Sterile water in volume equal to that of the comparator drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin E — A single intragastric dose of dl-α-tocopheryl acetate 50 IU/kg.
  Other Names: Aquasol E®
  Arms: Vitamin E
Drug: Placebo — Sterile water in volume equal to that of the comparator drug
  Arms: Placebo

SUMMARY:
The purpose of this pilot trial is to test the safety and efficacy of administering one dose of vitamin E, via a tube into the stomach, to extremely preterm infants (less than 27 weeks gestation and less than 1000 grams birth weight). This pilot will examine whether a single dose of vitamin E will be absorbed into the infants' bloodstreams with resulting serum α-tocopherol level in the target range of 1-3 mg/dl.

DETAILED DESCRIPTION:
Intraventricular hemorrhage (IVH) -- bleeding into the brain's ventricular system -- is one of the most common complications of prematurity, affecting an estimated 10-40% of very low birth weight (<1500 g) infants born at less than 35 weeks of gestation. Mortality from severe (high-grade) IVH is 27-50%. Severe IVH can result in developmental delays and life-long neurological deficits, including cerebral palsy and seizures.

A number of strategies have been used in efforts to prevent IVH, including: antenatal corticosteroids, maternal vitamin K, delayed clamping of the umbilical cord, indomethacin, ethamsylate, inositol, and muscle paralysis. With the exception of antenatal corticosteroids and indomethacin, these measures have met with only limited success. Supplemental vitamin E, given in the first few hours of life to all premature infants, offers a promising low-risk approach to preventing and/or lessening the severity of IVH.

This safety and efficacy pilot trial will examine whether one dose of vitamin E (dl-α-tocopheryl acetate), given intragastrically to preterm infants <27 weeks gestation and <1000 grams birth weight, will produce blood serum α-tocopherol levels in the target range of 1-3 mg/dl. Based on the results of this pilot, a Phase III randomized control trial will be developed to test whether a single dose of vitamin E can reduce the incidence of death or neurodevelopmental impairment at 18-22 months corrected age in these preterm infants.

Most intraventricular hemorrhages occur in the first 72 hours after birth. Because of this, to prevent IVH, it must be given as soon as possible after birth. Eligible, consented infants will be assigned to either a vitamin E group or a placebo group. Infants in the vitamin E group will receive 1.0 ml/kg of dl-α-tocopheryl acetate (Aquasol E®); infants in the placebo control group will receive a similar amount of sterile water. The dose will be given within 4 hours of birth via a tube into the stomach. Blood samples will be taken from all infants before the dose is given, 24 hours after dosing, and 7 days after dosing to measure how well the vitamin E is absorbed into the bloodstream.

ELIGIBILITY:
Inclusion Criteria:

* Less than 27 completed weeks gestational age
* Birth weight less than 1,000 grams
* Inborn infants

Exclusion Criteria:

* Infant's treatment will be limited based on poor prognosis
* Umbilical cord or blood pH below 7.0
* Antenatally diagnosed brain abnormality, including hemorrhage
* Major congenital malformations, including those for which feeding is contraindicated
* Mother of infant enrolled in a clinical trial of vitamin E supplementation
* Mother of infant reports self administration of monovitamin supplements of vitamin E during pregnancy or labor
* Infant has received supplemental vitamin E (except multivitamin additive in parenteral nutrition or through enteral milk or formula feeds)
* Greater than four hours of age

Max Age: 4 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Serum tocopherol levels | Birth to 7 days
  Blood samples will be tested for tocopherol levels at baseline, 24 hours, and 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Abbot R. Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Michele C. Walsh, MD MS, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Ronald N. Goldberg, MD, Principal Investigator — Duke University; Barbara J. Stoll, MD, Principal Investigator — Emory University; Brenda B. Poindexter, MD MS, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P. Van Meurs, MD, Principal Investigator — Stanford University; Ivan D. Frantz, III, MD, Principal Investigator — Tufts Medical Center; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Edward F. Bell, MD, Study Chair — University of Iowa; Kristi L. Watterberg, MD, Principal Investigator — University of New Mexico; Pablo J. Sanchez, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Kathleen A. Kennedy, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Roger G. Faix, MD, Principal Investigator — University of Utah; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Result] Bell EF, Hansen NI, Brion LP, Ehrenkranz RA, Kennedy KA, Walsh MC, Shankaran S, Acarregui MJ, Johnson KJ, Hale EC, Messina LA, Crawford MM, Laptook AR, Goldberg RN, Van Meurs KP, Carlo WA, Poindexter BB, Faix RG, Carlton DP, Watterberg KL, Ellsbury DL, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Serum tocopherol levels in very preterm infants after a single dose of vitamin E at birth. Pediatrics. 2013 Dec;132(6):e1626-33. doi: 10.1542/peds.2013-1684. Epub 2013 Nov 11. PMID 24218460
- See also: Neonatal Research Network website — http://neonatal.rti.org